CLINICAL TRIAL: NCT00064376
Title: A Phase II Trial Of Paricalcitol In Myelodysplastic Syndromes
Brief Title: Paricalcitol in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, H. Phillip Koeffler, Director, Medicine / Hematology/Oncology, Cedars-Sinai Medical Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000315451; CSMC-IRB-4107-01
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic | interventions — paricalcitol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: paricalcitol

SUMMARY:
RATIONALE: Paricalcitol is a form of vitamin D that may help myelodysplastic cells develop into normal bone marrow cells.

PURPOSE: Phase II trial to study the effectiveness of paricalcitol in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical effects of paricalcitol in patients with myelodysplastic syndromes.
* Determine whether this drug can improve RBC, WBC, or platelet counts in these patients.
* Determine whether this drug can decrease the risk of development of leukemia without causing undue toxicity in these patients.

OUTLINE: Patients receive oral paricalcitol daily for 4 months in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical diagnosis of myelodysplastic syndromes according to the modified FAB classification

  * Confirmed by bone marrow aspiration showing blast and promyelocyte count no greater than 30% of the bone marrow differential
* Patients with refractory anemia with ringed sideroblasts are eligible provided there was no response to a 3-week course of prior high-dose pyridoxine

PATIENT CHARACTERISTICS:

Age

* 25 to 100

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 2.0 mg/dL

Renal

* Creatinine less than 2.5 mg/dL
* Calcium normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior sensitivity to paricalcitol or any component of its formulation
* No prior cholecalciferol toxicity
* No other concurrent acute illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 5 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 5 weeks since prior radiotherapy

Surgery

* Prior recent surgery allowed, if fully recovered

Other

* More than 5 weeks since prior megadose vitamins
* No concurrent cholecalciferol, phosphate, calcium, or cholestyramine
* No concurrent digoxin

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05 (Actual); Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Phillip Koeffler, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California, United States